CLINICAL TRIAL: NCT02681666
Title: A Pilot, Randomized Trial of Mindfulness-based Irritable Bowel Syndrome Eating Awareness Training as Compared to the Standard Low Fermentable Oligosaccharide, Disaccharide, Monosaccharide and Polyol Diet in Patients With IBS
Brief Title: Mindfulness-Based Eating in Patients With Irritable Bowel Syndrome
Acronym: MB-IBS-EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Daniel A. Sussman, MD, MSPH, Associate Professor of Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150591
Record Dates: First submitted 2015-08-17; First posted 2016-02-12 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Abdominal Pain; Irritable Bowel Syndrome; IBS
Keywords: FODMAP Diet; Bowel Habit; Rome IV Criteria; Mindfulness; Abdominal pain; Irritable Bowel Syndrome
MeSH Terms: conditions — Abdominal Pain; Irritable Bowel Syndrome | interventions — Diet Therapy; FODMAP Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FODMAPs CONTROL arm (Active Comparator): Dietary intervention in this cohort with irritable bowel syndrome will be administered a low Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols diet by a dietician.
  Interventions: Dietary Supplement: Dietary intervention
- MB-IBS-EAT INTERVENTION STUDY arm (Experimental): Irritable Bowel Syndrome eating awareness training intervention will be started in a comprehensive 8 weekly sessions of Mindfulness eating training.
  Interventions: Behavioral: Irritable Bowel Syndrome eating awareness training

INTERVENTIONS:
Dietary Supplement: Dietary intervention — Sessions will be spent with patients discussing the FODMAPs (fermentable oligosaccharides, disaccharides, monosaccharides, and polyols) diet and how to use this diet to treat their Irritable Bowel Syndrome.
  Other Names: FODMAPs Diet
  Arms: FODMAPs CONTROL arm
Behavioral: Irritable Bowel Syndrome eating awareness training — A type of meditation about their eating habits.
  Other Names: MB-IBS-EAT
  Arms: MB-IBS-EAT INTERVENTION STUDY arm

SUMMARY:
This pilot study will be a randomized parallel trial comparing Mindfulness-Based Irritable Bowel Syndrome Eating Awareness Training done over an 8 week period to a standard low Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols diet.

DETAILED DESCRIPTION:
This study is supported by findings that Irritable Bowel Syndrome patients have an alteration of the hypothalamus-pituitary-adrenal stress axis such that cortisol levels are elevated. Stress-induced release of corticotropin-releasing factor alters gastric digestion and gastrointestinal motility. Furthermore, stress is a contributing factor to the immune activation and low-grade inflammation observed in Irritable Bowel Syndrome with overall physical and psychological distress correlating with percentage of activated natural killer and T cells. In addition, the brain-gut axis is a proposed mechanism in Irritable Bowel Syndrome due to dysregulated enteric nervous system and central nervous system events. The central nervous system may perceive visceral stimuli from the gut mucosa when inflammation or injury causes afferent nerve sensitization.

Regardless of the specific pathophysiologic basis of Irritable Bowel Syndrome, the current aim of treatment is to improve quality of life, treatments include dietary alterations and psychological therapy such as cognitive behavioral therapy to aid symptomatic relief. The most common dietary intervention in patients with Irritable Bowel Syndrome is the fermentable oligosaccharide, disaccharide, monosaccharide and polyol restricted diet. However, adherence to this diet is very difficult with most patients with Irritable Bowel Syndrome failing to continue eliminating foods leading to bloating or pain. Various psychological therapies have been implemented in the past with the most successful of these being cognitive behavioral therapy. The beneficial results of incorporating mindfulness-based interventions to improve myriad health-related problems, such as Irritable Bowel Syndrome, anxiety disorders , psychological distress, quality of life, depression fibromyalgia , diabetes , and eating disorders has grown considerably in the recent past. Mindfulness Based Eating Awareness Training, which was developed based on Jon Kabat-Zinn's Mindfulness Based Stress Reduction program, has been shown to improve binge eating disorder and other food and stress-related problems. The effect of Mindfulness Based Eating Awareness Training is driven by the improved ability of practitioners to increase engagement in non-judgmental self-awareness behaviors designed to improve regulatory impulses and stress reactivity as well as to nurture awareness of emotional status and outside triggers. The investigators have developed a 12 week Mindfulness-Based Irritable Bowel Syndrome Eating Awareness Training inspired by relevant pieces of the Mindfulness Based Eating Awareness Training program. Mindfulness based interventions integrate moment by moment awareness of bodily sensations, observations, thoughts, and feelings while suspending judgments of self. Successful Irritable Bowel Syndrome treatment modalities have been elusive, but have a strong food and stress-reactive association making this medical condition ideal for a mindfulness treatment intervention. The usual diet for Irritable Bowel Syndrome is an elimination diet of fermentable carbohydrates (of varying sugar lengths) and polyols (sugar alcohols and stone fruits) called the Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols elimination diet. Patients with Irritable Bowel Syndrome who follow a Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols diet receive suboptimal nutrient intake over long time periods while attempting to discern which food groups are digestible and which others are intolerable, with mixed findings of improvement in quality of life, and other stress-related measures.

After eligibility is established, written informed consent will be obtained and randomization will be conducted to place participants in either the mindfulness-based Irritable Bowel Syndrome- eating awareness training group or the Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols group and pre-baseline testing will be performed on both groups. Two-four weeks later participants will receive baseline testing at their first session of both arms of the study. Four weeks later, participants in both study arms will receive a follow up assessment testing. Directly following the eight week intervention or Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols arm, participants will receive post-intervention testing 1.

At 2 and 4 weeks following the intervention or Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols FODMAPs) arm, post-intervention testing 2 and post-intervention testing 3 will take place, respectively for a total of 12 weeks.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged 18 and over
* Meet Rome III criteria for diagnosis of Irritable Bowel Syndrome
* Subjects with legal and mental capacity to understand and sign an informed consent.

Exclusion criteria: The following subjects will be excluded from the study:

* Pregnant patients
* Subjects with active malignancy in the previous five years
* Current or prior history of alcohol or drug abuse
* Any history of eating disorder such as anorexia or bulimia
* Subjects taking yoga or with prior history of mindfulness therapy within 3 months of enrolment
* Subjects currently on a FODMAP diet.
* Patients with psychiatric illnesses other than depression or anxiety disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2017-12-26 (Actual)

PRIMARY OUTCOMES:
Change in Global Improvement Scale score | Baseline, 4 weeks, 8 weeks, 12 weeks
  This questionnaire provides an overall assessment of how much a patient's symptoms and behaviors have improved or worsened since the start of treatment.

SECONDARY OUTCOMES:
Change in score of IBS-Quality of Life questionnaire | Baseline, 4 weeks, 8 weeks, 12 weeks
  This questionnaire is a 34-item instrument developed and validated for measurement of health-related quality of life in non-subtyped IBS patients. [doi: 10.1186/1477-7525-11-208]
Change in score of Irritable Bowel Syndrome - Severity Scoring System | Baseline, 4 weeks, 8 weeks, 12 weeks
  "This scale evaluates primarily the intensity of IBS symptoms during a 10-day period: abdominal pain, distension, stool frequency and consistency, and interference with life in general. The IBS-SSS calculates the sum of these 5 items each scored on a visual analog scale from 0 to 100." [doi:10.1038/ajg.2011.201]
Change in score in Perceived Stress Scale | Baseline, 4 weeks, 8 weeks, 12 weeks
  This questionnaire measures the degree to which situations in one's life are appraised as stressful.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sussman, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided